CLINICAL TRIAL: NCT05449717
Title: A Prospective Cohort Study on the Incidence of Relapse and Post-Kala-Azar Dermal Leishmaniasis After Treatment for Primary Visceral Leishmaniasis in South Sudan
Brief Title: Incidence of Relapse and Post-Kala-Azar Dermal Leishmaniasis in South Sudan
Acronym: PKDL
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Drugs for Neglected Diseases (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: PKDL/2184
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Leishmaniasis; Leishmaniasis, Visceral; Post-kala-azar Dermal Leishmaniasis
Keywords: Leishmaniasis; Leishmaniasis, Visceral; Post-Kala-Azar Dermal Leishmaniasis; South Sudan; Kala-Azar
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Visceral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to describe the burden of Post-Kala-Azar Dermal Leishmaniasis and visceral leishmaniasis relapse in a cohort of patients discharged after successful treatment of primary visceral leishmaniasis.

DETAILED DESCRIPTION:
This prospective, observational cohort study aims to describe the burden of Post-Kala-Azar Dermal Leishmaniasis and visceral leishmaniasis relapse in a cohort of patients discharged after successful treatment of primary visceral leishmaniasis from a hospital in Lankien, South Sudan.

ELIGIBILITY:
Inclusion Criteria:

* Primary visceral leishmaniasis patients who had a confirmed (serological and/or parasitological) diagnosis at admission, and who were discharged after successful treatment
* Availability for follow up visits
* Provision of informed consent, and in the case of minors 12 to 17 years of age, assent as well

Exclusion Criteria:

* Unavailability for follow-up visits due to distance, inaccessibility, or refusal to participate
* Diagnosis of prior primary visceral leishmaniasis done only on clinical basis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Successfully treated and discharged primary cases of visceral leishmaniasis from the Médecins Sans Frontières-Operational Center Amsterdam (MSF-OCA)-run hospital in Jonglei State, South Sudan
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Incidence of post-kala-azar-dermal leishmaniasis (PKDL) | 12 months
  To determine the incidence of PDKL after initial successful treatment of primary visceral leishmaniasis (VL) over a period of 12 months
Incidence of VL relapse | 12 months
  To determine the incidence of VL relapse after initial successful treatment of primary VL over a period of 12 months

SECONDARY OUTCOMES:
Time of onset of visceral leishmaniasis (VL) relapse or post-kala-azar-dermal leishmaniasis (PKDL) | 12 months
  To determine the time of onset of VL relapse or PKDL at follow-up 1, 3, 6, 9, and 12 months after initial successful treatment of primary VL
Characterize PKDL lesions | 12 months
  To characterize (e.g., grade, distribution) PKDL lesions
Risk factors for the development of VL relapse or PKDL | 12 months
  To assess the risk factors for the development of VL relapse or PKDL after initial successful treatment of primary VL
Rate and time period to self-healing of PKDL | 12 months
  To determine the rate and time period to self-healing of PKDL

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Coulborn, MPH, Principal Investigator — Epicentre; Margriet den Boer, MD, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (1):
- Lankien Hospital, Lankien, Jonglei, South Sudan

IPD SHARING:
Plan to Share IPD: Yes
A long-standing individual participant data (IPD) sharing plan already exists between Epicentre and Médecins Sans Frontières.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be shared as they become available, for the duration of the project, estimated at 3 years.
Access Criteria: Existing co-investigator, or permission of Co-Principal Investigators, on research protocol.